CLINICAL TRIAL: NCT00766194
Title: Nasopharyngeal Pressure Measurement During Neonatal Nasal Respiratory Support
Status: Terminated | Type: Observational
Why Stopped: slow enrollment
Sponsor: University of Utah (Other)
Responsible Party: Don Null M.D., Unviersity of Utah Pediatrics / Neonatology
Other Study IDs: 22939/36001
Record Dates: First submitted 2008-09-03; First posted 2008-10-03 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Nasopharyngeal Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will measure nasopharyngeal pressure in neonates using a miniature high resolution catheter-tip pressure transducer. Any neonatal intensive care patient being treated with nasal respiratory support (e.g., nasal continuous positive airway pressure, nasal cannula flow either high (>1 LPM) or low (<1 LPM), and nasal prong ventilation either intermittent mandatory or high-frequency) will be eligible for study. The catheter-tip transducer will be placed within a standard gavage feeding tube catheter and introduced through the mouth into the posterior nasopharynx where continuous measurements will be made over 15 minutes. The 15 minute recording will be divided into 5 three minute segments, including a baseline recording at the ordered settings of pressure or flow, a recording at 1 level above baseline, a recording back at baseline, a recording 1 level below baseline, and a final segment back at baseline. The order of increase-decrease or decrease-increase from baseline will be by random sequence. Measurements may be repeated with any change in nasal gas flow or pressure ordered for patient care. These measurements will be used to correlate the ordered nasal respiratory support therapy with the actual upper airway pressure created by the therapy.

DETAILED DESCRIPTION:
Non-invasive respiratory treatments are being used more frequently during neonatal intensive care. High-flow nasal cannula,1-2 nasal continuous positive airway pressure,3 nasal intermittent mandatory or synchronized ventilation,4 and high-frequency nasal continuous airway pressure5-6 are some of these modalities. These non-invasive therapies attempt to provide adequate oxygen delivery, positive end-expiratory pressure to maintain lung recruitment, and ventilation assistance without the need for endotracheal intubation. The benefits may be substantial, including decreased frequency of nosocomial infection, decreased risk for lung injury, and prevention of arrest in pulmonary development for those very preterm infants with immature lungs. However, there are very few reports of actual measurement of nasopharyngeal pressure during use of these non-invasive therapies.1,7 Combined, only 27 patients are included in two studies. Only one modality, high-flow nasal cannula, was evaluated. One study in 11 patients suggests a 2-3 cmH2O pressure drop exists between applied and delivered airway pressure.7 In order to better understand the relationship between applied and delivered airway pressures with all types of non-invasive therapy, we propose to measure nasopharyngeal pressure in neonates being treated with these modes of respiratory support.

If non-invasive respiratory support is initiated as part of routine pulmonary therapy for a neonate admitted to neonatal intensive care, the infant will be considered eligible for study if no exclusion criteria are met. Informed consent/parental permission will be requested and if obtained, the infant will be included for study.

The study procedure will be as follows:

* Care information will be documented, to include the infant's post-menstrual and post-delivery age, current weight, current level of supplemental oxygen administration, current pulse oximeter saturation level, applied flow and pressure settings, and if non-invasive ventilation is being used, the ventilator parameters.
* A high resolution fiber optic pressure tip transducer catheter will be inserted into a 5F or similar size fenestrated tube (such as an Anderson catheter) and introduced through the mouth towards the posterior pharynx. The pressure transducer/catheter combination will only be inserted the minimum distance to obtain a stable pressure signal reading and not produce choking or gagging in the infant. If the infant demonstrates choking or gagging, the tube will be withdrawn to a position that does not produce choking or gagging in the infant. If the pressure signal suggests that the catheter openings may be occluded with mucous, 5mL of air may be injected into the catheter to clear the mucous and obtain a satisfactory recording.
* A 1 to 5 minute recording will be made from the pressure transducer onto a notebook computer at the current non-invasive therapy settings.
* Two more 1 to 5 minute recordings will be made, either 0.5-1.0 cmH2O or 0.5-1.0 liter per minute flow (depending on the non-invasive modality) above and below the current settings. The order of the increase or decrease will be by random sequence.
* A final fourth 1 to 5 minute recording will be made when the settings have been returned to the current baseline settings.
* Pulse oximeter saturation will be recorded both before and after each recording.
* A study infant will undergo a baseline study procedure, and re-studied whenever the non-invasive therapy settings are changed based on clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Any infant admitted to neonatal intensive care who is treated with a modality of non-invasive respiratory support, such as low or high flow nasal cannula; nasal prong, catheter or mask continuous distending pressure; or nasal ventilation either intermittent mandatory, synchronized or high frequency will be eligible for study.

Exclusion Criteria:

* Patients with oral, nasal, or palatal deformities who can not otherwise be fitted with cannula or mask will be excluded from the study.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any infant admitted to neonatal intensive care who is treated with a modality of non-invasive respiratory support, such as low or high flow nasal cannula; nasal prong, catheter or mask continuous distending pressure; or nasal ventilation either intermittent mandatory, synchronized or high frequency will be eligible for study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald .Null, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah / Primary Childrens Medical Center, Salt Lake City, Utah, United States